CLINICAL TRIAL: NCT02802033
Title: DegenPRO: A Multicenter Prospective Registry for the Management of Degenerative Spine Disorders
Brief Title: A Multicenter Prospective Registry for the Management of Degenerative Spine Disorders
Status: Active, not recruiting | Type: Observational
Sponsor: AO Innovation Translation Center (Other)
Collaborators: AO Foundation, AO Spine (Other)
Responsible Party: Sponsor
Other Study IDs: DegenPRO
Record Dates: First submitted 2016-05-27; First posted 2016-06-16 (Estimated); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Degenerative Diseases, Spinal Cord
Keywords: Registry; Spine; Osteobiologics; Spinal Fusion
MeSH Terms: conditions — Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Details regarding the degenerative spine disorders will be collected with a specific focus on the use of osteobiologics in treating degenerative conditions and their impact on fusion, as well as patient-reported outcomes for these conditions.

DETAILED DESCRIPTION:
The registry is designed to be open-ended. However, a statistical evaluation of the content und structure of database and CRFs in order to investigate the feasibility and quality of data collection is planned to take place prior to the registry expansion.

Variables applicable to patients with a degenerative spine disorder which will be collected in the registry include:

* Patient details
* Symptoms
* Diagnosis
* Imaging assessment
* Treatment details

Feasibility phase:

The statistical evaluation of the feasibility and quality of data collection will be performed after the first 5 sites have each enrolled 12 patients with a degenerative pathology and documented one follow-up visit. During this evaluation, enrolment of further patients can be continued.

Based on the findings of this feasibility phase, adjustments to the existing database can be performed before the registry is rolled out on larger scale.

Registry expansion:

Following the evaluation process of the feasibility phase, the registry will be expanded to allow data entry in more sites globally. Multi-site participation of this registry will be rolled-out in stages, and will be offered to sites with appropriate expertise which are selected based on their potential (interest, resources and expected patient volume).

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older
* Patient diagnosed with a degenerative spine disorder who receives treatment for the degenerative spine disorder
* Patient capable of understanding the content of the patient information / Informed Consent Form
* Patient willing and able to participate in the registry
* Patient who has agreed to participate in the registry by providing consent according to the applicable local law and the declaration of Helsinki

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a degenerative spine disorder
Sampling Method: Non-Probability Sample
Enrollment: 908 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Use of Osteobiologics - Within the registry information on the use of osteobiologis (autografts, allografts, BMA/cells, BMP, DBM, matrices/carriers, platelets) are collected | Every standard of care scheduled follow-up visit up to 3 years
  Osteobiologics are classified as autogenous bone graft substitutes, extenders, or enhancers. Types of osteobiologics include demineralized bone matrices (DBM), allografts and allograft formulations, synthetic bone grafts, bone morphogenic proteins, bone marrow aspirate systems, stem cells and platelet-rich plasma systems. The biologics are generally defined as being derived from or replicating natural substances. The osteobiologics are defined as such by possessing one or more of the following properties: osteoinductivity, osteoconductivity, and osteogenicity. Although biologics are classically defined as being derived from or replicating natural substances, a broader definition of an osteobiologic includes synthetic derivatives that may not replicate natural substances, but serve as a bone graft substitute, extender or enhancer.
  There is not yet defined how the data will be analysed. Data collected can help drive hypotheses and might help to answer unforeseen questions over time.

SECONDARY OUTCOMES:
Neck, Arm, Back, Leg, Thoracic pain Numeric Rating Scale (NRS) | Every standard of care scheduled follow-up visit up to 3 years
Neck Disability Index (NDI) | Every standard of care scheduled follow-up visit up to 3 years
Oswestry Disability Index (ODI) | Every standard of care scheduled follow-up visit up to 3 years
Euroqol EQ-5D-3L | Every standard of care scheduled follow-up visit up to 3 years
Short Form (SF)-36 V2 | Every standard of care scheduled follow-up visit up to 3 years
Modified Zung Depression Index | Every standard of care scheduled follow-up visit up to 3 years
Distress and Risk Assessment Method (DRAM) | Every standard of care scheduled follow-up visit up to 3 years
Scoliosis Research Society (SRS)-22 Questionnaire | Every standard of care scheduled follow-up visit up to 3 years
Modified Japanese Orthopedic Association Score (mJOA) | Every standard of care scheduled follow-up visit up to 3 years
Type of fusion that was performed (posterior and/or anterior/interbody fusion) | 6 months after surgery, if this time point is collected as per standard of care
  Data will be entered in the database but there is not yet defined how the data will be analysed. Data collected can help drive hypotheses and might help to answer unforeseen questions over time.
Type of fusion that was performed (posterior and/or anterior/interbody fusion) | 12 months after surgery, if this time point is collected as per standard of care
  Data will be entered in the database but there is not yet defined how the data will be analysed. Data collected can help drive hypotheses and might help to answer unforeseen questions over time.
Fusion: Bridging trabecular bone across the segment, bone graft resorption, implant subsidence/migration, fatigue failure of spinal instrumentation, radioluciencies around screws, instability on flexion/extension views | 6 months after surgery, if this time point is collected as per standard of care
  Radiological source for interpretation (Clinical assessment, radiographs, CT, MRI, bone scan, other) Data will be entered in the database but there is not yet defined how the data will be analysed. Data collected can help drive hypotheses and might help to answer unforeseen questions over time.
Fusion: Bridging trabecular bone across the segment, bone graft resorption, implant subsidence/migration, fatigue failure of spinal instrumentation, radioluciencies around screws, instability on flexion/extension views | 12 months after surgery, if this time point is collected as per standard of care
  Radiological source for interpretation (Clinical assessment, radiographs, CT, MRI, bone scan, other) Data will be entered in the database but there is not yet defined how the data will be analysed. Data collected can help drive hypotheses and might help to answer unforeseen questions over time.
Success of fusion | 6 months after surgery, if this time point is collected as per standard of care
  Data will be entered in the database but there is not yet defined how the data will be analysed. Data collected can help drive hypotheses and might help to answer unforeseen questions over time.
Success of fusion | 12 months after surgery, if this time point is collected as per standard of care
  Data will be entered in the database but there is not yet defined how the data will be analysed. Data collected can help drive hypotheses and might help to answer unforeseen questions over time.

OTHER OUTCOMES:
Information on postoperative adverse events | Every standard of care scheduled follow-up visit up to 3 years
  Data will be entered in the database but there is not yet defined how the data will be analysed. Data collected can help drive hypotheses and might help to answer unforeseen questions over time.
Duration of postoperative adverse event | Every standard of care scheduled follow-up visit up to 3 years
  Data will be entered in the database but there is not yet defined how the data will be analysed. Data collected can help drive hypotheses and might help to answer unforeseen questions over time.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Yoon, MD, Principal Investigator — Principal Coordinating Investigator
Locations (7):
- United States (5):
  - USC Spine Center, Keck Medical Center of USC, Los Angeles, California
  - Emory University School of Medicine, Atlanta, Georgia
  - The Johns Hopkins University, Baltimore, Maryland
  - Mount Sinai Hospital, New York, New York
  - New York Presbyterian - Columbia University Medical Center, New York, New York
- BG-Clinic Bergmannstrost, Halle, Germany
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No